CLINICAL TRIAL: NCT00257777
Title: Intermittent Cold Blood vs Crystalloid Cardioplegia in Aortic Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVR03; AVR03
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2005-11

CONDITIONS: Aortic Valve Disease; Coronary Artery Disease
MeSH Terms: conditions — Aortic Valve Disease; Coronary Artery Disease

INTERVENTIONS:
Procedure: Myocardial protection techniques

SUMMARY:
Controversies still exists concerning the overall clinical effects of blood-based vs. crystalloid- based cardioplegic solution for myocardial protection during cardiac arrest. Both techniques are used world-wide. No larger prospectively randomized studies comparing the two methods have been reported. The aim of this study is to collect a large number of clinical data to create a proper basis for evaluation of the two techniques.

DETAILED DESCRIPTION:
All patients admitted for aortic valve replacement with or without concomitant CABG and operated by E.Ø. or G.T. are included in the study. All preoperative, operative and postoperative data are prospectively recorded, focusing on clinical outcome parameters

ELIGIBILITY:
Aortic valve replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2003-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Myocardial function,
postoperative ventilatory support, postoperative arrhythmia,
blood transfusions,
physical recovery,
mortality.

SECONDARY OUTCOMES:
Costs

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Øvrum, MD,PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- RRHF, Oslo, Norway